CLINICAL TRIAL: NCT00560391
Title: A Phase I Single Arm Dose Escalation Study of the Combination of Dasatinib (Sprycel®) With Lenalidomide (Revlimid®) and Dexamethasone in Subjects With Relapsed and/ or Refractory Multiple Myeloma
Brief Title: Dasatinib in Combination With Revlimid (and Dexamethasone)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-180
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dasatinib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dasatinib, 70 mg + Lenalidomide, 15 mg + Dexamethasone, 40 mg (Experimental): Participants received a combination of dasatinib, 70 mg QD, lenalidomide, 15 mg QD, and dexamethasone, 40 mg QD, weekly on Days 1, 8, 15, and 22, in 28-day cycles.
  Interventions: Drug: Dasatinib, 70 mg + Lenalidomide, 15 mg + Dexamethasone, 40 mg
- Dasatinib, 70 mg + Lenalidomide, 20 mg + Dexamethasone, 40 mg (Experimental): Participants received a combination of dasatinib, 70 mg QD, lenalidomide, 20 mg QD, and dexamethasone, 40 mg QD, weekly on Days 1, 8, 15, and 22, in 28-day cycles.
  Interventions: Drug: Dasatinib, 70 mg + Lenalidomide, 20 mg + Dexamethasone, 40 mg
- Dasatinib, 100 mg + Lenalidomide, 20 mg + Dexamethasone, 40 mg (Experimental): Participants received a combination of dasatinib, 100 mg QD, lenalidomide, 20 mg QD, and dexamethasone, 40 mg QD, weekly on Days 1, 8, 15, and 22, in 28-day cycles.
  Interventions: Drug: Dasatinib, 100 mg + Lenalidomide, 20 mg + Dexamethasone, 40 mg
- Dasatinib, 100 mg + Lenalidomide, 25 mg + Dexamethasone, 40 mg (Experimental): Participants received a combination of dasatinib, 100 mg QD, lenalidomide, 25 mg QD, and dexamethasone, 40 mg QD, weekly on Days 1, 8, 15, and 22, in 28-day cycles.
  Interventions: Drug: Dasatinib, 100 mg + Lenalidomide, 25 mg + Dexamethasone, 40 mg
- Dasatinib, 140 mg + Lenalidomide, 25 mg + Dexamethasone, 40 mg (Experimental): Participants received a combination of dasatinib, lenalidomide, and dexamethasone in varying doses in 28-day cycles.
  Interventions: Drug: Dasatinib, 140 mg + Lenalidomide, 25 mg + Dexamethasone, 40 mg

INTERVENTIONS:
Drug: Dasatinib, 70 mg + Lenalidomide, 15 mg + Dexamethasone, 40 mg — Participants received dasatinib, 70 mg once daily (QD), for 28 days plus lenalidomide, 15 mg QD, for 21 days plus dexamethasone, 40 mg QD, weekly on Days 1, 8, 15, and 22.
  Other Names: Sprycel®; BMS-354825; Revlimid®
  Arms: Dasatinib, 70 mg + Lenalidomide, 15 mg + Dexamethasone, 40 mg
Drug: Dasatinib, 70 mg + Lenalidomide, 20 mg + Dexamethasone, 40 mg — Participants received dasatinib, 70 mg QD, for 28 days plus lenalidomide, 20 mg QD, for 21 days, plus dexamethasone, 40 mg QD, weekly on Days 1, 8, 15, and 22.
  Other Names: Sprycel®; BMS-354825; Revlimid®
  Arms: Dasatinib, 70 mg + Lenalidomide, 20 mg + Dexamethasone, 40 mg
Drug: Dasatinib, 100 mg + Lenalidomide, 20 mg + Dexamethasone, 40 mg — Participants received dasatinib, 100 mg QD, for 28 days, plus lenalidomide, 20 mg QD, for 21 days, plus dexamethasone, 40 mg QD, weekly on Days 1, 8, 15, and 22.
  Other Names: Sprycel®; BMS-354825; Revlimid®
  Arms: Dasatinib, 100 mg + Lenalidomide, 20 mg + Dexamethasone, 40 mg
Drug: Dasatinib, 100 mg + Lenalidomide, 25 mg + Dexamethasone, 40 mg — Participants received dasatinib, 100 mg QD, for 28 days, plus lenalidomide, 25 mg QD, for 21 days, plus dexamethasone, 40 mg QD, weekly on Days 1, 8, 15, and 22.
  Other Names: Sprycel®; BMS-354825; Revlimid®
  Arms: Dasatinib, 100 mg + Lenalidomide, 25 mg + Dexamethasone, 40 mg
Drug: Dasatinib, 140 mg + Lenalidomide, 25 mg + Dexamethasone, 40 mg — Participants received dasatinib, 140 mg QD, for 28 days, plus lenalidomide, 25 mg QD, for 21 days, plus dexamethasone, 40 mg QD, weekly on Days 1, 8, 15, and 22. Cohort includes 4 participants who received treatment during the dose-finding phase and 13 participants who received treatment in the dose-expansion phase.
  Other Names: Sprycel®; BMS-354825; Revlimid®
  Arms: Dasatinib, 140 mg + Lenalidomide, 25 mg + Dexamethasone, 40 mg

SUMMARY:
The purpose of this study was to determine the safety and tolerability of dasatinib when given in combination with lenalidomide and a low dose dexamethasone for the treatment of relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Men and women age ≥ 18 years
* Confirmed diagnosis of multiple myeloma (MM) with measurable disease assessed within 1 month prior to treatment initiation
* Evidence of relapsed or refractory disease and at least one prior therapy for MM
* Eastern Cooperative Oncology Group Scale (ECOG) Performance Status of 0 - 2
* Last MM treatment at least 21 days prior to treatment initiation• Bone marrow transplant (BMT) at least 3 months prior to treatment initiation
* Required baseline hematology and chemistry parameters
* Resolution of acute toxicity due to prior therapy to Grade <2 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Men whose sexual partners are women of child bearing potential (WOCBP) or WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least one month (4 weeks) before and for at least one month (4 weeks) after the last dose of study medication.
* Clinically significant cardiac disease (New York Heart Association [NYHA] Class III or IV)
* Abnormal corrected QT interval using Fridericia's formula (QTcF) interval prolonged (> 450 msec)
* Medications that are generally considered to have a risk of causing "Torsades de Pointes"
* Malabsorption syndrome or uncontrolled gastrointestinal toxicities
* Clinically significant pleural effusion in the previous 12 months or current ascites
* Clinically-significant coagulation or platelet function disorder
* Dementia, chronic medical or psychiatric condition, or laboratory abnormality
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality, serious uncontrolled medical disorder or active infection
* Intolerance to dasatinib and/or lenalidomide
* Subjects with a history of severe rash, hypersensitivity reaction or anaphylaxis related to prior thalidomide treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States
- Local Institution, Prahran, Victoria, Australia
- France (2):
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 39 participants were enrolled in this study, 4 never received treatment due to screening failure. A total of 35 participants received treatment.
Groups:
- Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg: Participants were treated with a combination of dasatinib, lenalidomide and dexamethasone in 28 day cycles (dasatinib 70 mg QD for 28 days and lenalidomide 15 mg QD for 21 days, along with 40 mg QD of dexamethasone given weekly on Days 1, 8, 15, and 22).
- Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg: Participants were treated with a combination of dasatinib, lenalidomide and dexamethasone in 28 day cycles (dasatinib 70 mg QD for 28 days and lenalidomide 20 mg QD for 21 days, along with 40 mg QD of dexamethasone given weekly on Days 1, 8, 15, and 22).
- Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg: Participants were treated with a combination of dasatinib, lenalidomide and dexamethasone in 28 day cycles (dasatinib 100 mg QD for 28 days and lenalidomide 20 mg QD for 21 days, along with 40 mg QD of dexamethasone given weekly on Days 1, 8, 15, and 22).
- Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg: Participants were treated with a combination of dasatinib, lenalidomide and dexamethasone in 28 day cycles (dasatinib 100 mg QD for 28 days and lenalidomide 25 mg QD for 21 days, along with 40 mg QD of dexamethasone given weekly on Days 1, 8, 15, and 22).
- Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg: Participants were treated with a combination of dasatinib, lenalidomide and dexamethasone in 28 day cycles (dasatinib 140 mg QD for 28 days and lenalidomide 25 mg QD for 21 days, along with 40 mg QD of dexamethasone given weekly on Days 1, 8, 15, and 22). Cohort includes 4 participants treated for dose -finding phase and 13 participants treated in dose expansion phase.
Period: Overall Study
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Started | 6 (Participants who received treatment) | 3 (Participants who received treatment) | 3 (Participants who received treatment) | 6 (Participants who received treatment) | 17 (Participants who received treatment)
Completed | 6 (Completed=off treatment;Disease progression-1;Death-1;Max. clinical benefit-2;Study drug toxicity-2) | 3 (Completed=off treatment; Disease progression-1;Death-1; Unrelated AE-1) | 3 (Completed=off treatment; Disease progression-1;Maximum clinical benefit-1; Unrelated AE-1) | 5 (Completed=off treatment; Disease progression-2; Unrelated AE 1 and Subject request 2) | 15 (Completed=offtreatment;Disease progression-6;Study drug toxicity-7; Unrelated AE-1,Subject request-1)
Not Completed | 0 | 0 | 0 | 1 | 2
Not completed — Still on treatment | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Total
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (11.75) | 69.3 (4.73) | 63.0 (11.14) | 69.7 (5.92) | 59.3 (8.06) | 63.4 (9.19)
Age, Customized [Number; unit: participants]
  21 - 45 years | 0 | 0 | 0 | 0 | 1 | 1
  46 - 65 years | 3 | 1 | 2 | 1 | 13 | 20
  66 - 75 years | 1 | 2 | 1 | 5 | 3 | 12
  >75 years | 2 | 0 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 4 | 7 | 18
  Male | 2 | 1 | 2 | 2 | 10 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 3 | 3 | 6 | 16 | 34
  Asian | 0 | 0 | 0 | 0 | 1 | 1
International Staging System (ISS) [Number; unit: participants] — The ISS is an updated staging system for multiple myeloma. ISS divides multiple myeloma into three stages, which indicate the effect the disease is having on the body and how quickly or slowly it may develop. The ISS is based on the levels of blood proteins beta-2 microglobulin (β2M) and albumin. Stage I= β2M: <3.5 mg/L, albumin: >=3.5 g/dL; Stage II= β2M level: < 3.5 mg/L and albumin: < 3.5 g/dL, or β2M =3.5 to 5.5 mg/dL; Stage III: β2M level: >=5.5 mg/L.
  participants
    Stage I | 1 | 0 | 1 | 0 | 4 | 6
    Stage II | 1 | 0 | 0 | 3 | 2 | 6
    Stage III | 1 | 2 | 0 | 1 | 1 | 5
    Not assessed | 3 | 1 | 2 | 2 | 10 | 18
Durie-Salmon Staging System [Number; unit: participants] — Myeloma is classified into 3 stages. Stage I: hemoglobin (Hb) >10g/dL, normal calcium levels, normal skeletal survey or single plasmacytoma or osteoporosis, serum paraprotein level<5g/dL if immunoglobulin G(IgG), <3g/dL if IgA, urinary light chain excretion<4g/24h. Stage II: fulfilling the criteria of neither I nor III. Stage III: Hb<8.5g/dL, high calcium >12mg/dL, Skeletal survey of 3 or more lytic bone lesions, serum paraprotein >7g/dL if IgG,>5g/dL if IgA, urinary light chain excretion >12g/24h. Each stage further subdivided: A= serum creatinine <2mg/dL and B= serum creatinine >2mg/dL.
  participants
    Stage IA | 3 | 1 | 2 | 1 | 2 | 9
    Stage IB | 0 | 0 | 0 | 0 | 0 | 0
    Stage IIA | 0 | 0 | 1 | 3 | 3 | 7
    Stage IIB | 0 | 0 | 0 | 0 | 0 | 0
    Stage IIIA | 3 | 2 | 0 | 0 | 6 | 11
    Stage IIIB | 0 | 0 | 0 | 0 | 0 | 0
    Not Assessed | 0 | 0 | 0 | 2 | 6 | 8
Time from diagnosis to first dosing [Median (Full Range); unit: years] | 4.9 [2 to 18] | 4.0 [1 to 5] | 7.5 [7 to 11] | 5.2 [1 to 6] | 3.7 [1 to 16] | 4.4 [1 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (RP2D) of the Combination (Dasatinib + Lenalidomide + Dexamethasone)
Description: The RP2D was based on the MTD which was defined as the maximum combined dose producing dose limiting toxicity (DLT) in < 33% of participants treated at the individual dose levels in the combination. The MTD is considered the last dose level combination tested just below the maximum administered dose (MAD) level combination and for which DLTs were observed in less than or equal to 33% of participants during the escalation and expansion phase. If MTD was not reached Please refer to Outcome Measure 2 for the complete definition of DLT.
Time Frame: From the date of first dose to end of treatment (median duration of dasatinib treatment=5.2 months [range 0 to 33 months]).
Population: All treated participants, participants who received at least 1 dose of dasatinib.
Measure: Number; unit: mg
Groups:
- All Treated Participants: Participants were treated with a combination of dasatinib, lenalidomide and dexamethasone in 28 day cycles; dasatinib (70/100 mg)QD for 28 days, dexamethasone (40mg)given weekly on Days 1, 8, 15, and 22 and lenalidomide (15/20/25mg)QD for 21 days.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 35
mg
  RP2D of dasatinib in the combination | 140
  RP2D of lenalidomide in the combination | 25
  RP2D dexamethasone in the combination | 40

2. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT)
Description: DLTs: At least possibly drug-related AEs occurring during the first cycle of treatment and are:GR4 neutropenia >5 days/neutropenic fever;platelet count <10000mm^3 on >1 occasion;GR4 fatigue,or 2-point decline in ECOG performance status;>=GR3 nausea,diarrhea,and vomiting despite medical intervention;Any other clinically significant non-hematologic toxicity of >=GR3 considered not related to underlying MM;Any GR3/4 laboratory abnormality requiring hospitalization;dose interruption of either dasatinib and/or lenalidomide for >15 days due to any toxicity related to treatment with the combination.
Time Frame: From the date of first dose until at least 30 days after the last dose of study drug (median duration of dasatinib treatment=5.2 months [range 0 to 33 months]).
Population: All treated participants, participants who received at least 1 dose of dasatinib. (Participants included from Cohort 5 are those involved in the dose escalation phase only.)
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 4
participants | 1 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants in the Dose Escalation Phase Who Reached Maximum Tolerated Dose (MTD) of Dasatinib With Lenalidomide and Dexamethasone
Description: The MTD is considered the last dose level combination tested just below the maximum administered dose (MAD) level combination and for which DLTs were observed in less than 33% of participants during the escalation and expansion phase. Please refer to outcome 2 for the complete definition of DLT. If the MTD was not reached at the highest dose administered as defined by protocol, the highest dose (dasatinib 140 mg QD + lenalidomide 25 mg QD) administered was selected for the dose expansion phase of the study.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 4
participants | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Complete Response and Very Good Partial Response
Description: Response criteria were based on The International Uniform Response Criteria for Multiple Myeloma (with a slight modification). Complete response was achieved when there was negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow. Very good partial response was achieved when serum and urine M-component was detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-component plus urine M-component < 100 mg per 24 hour.
Time Frame: Baseline, At the end of the treatment period (median duration of dasatinib treatment=5.2 months [range 0 to 33 months]).
Population: All treated participants, participants who received at least 1 dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 17
participants
  Complete response | 0 | 0 | 0 | 0 | 0
  Very good partial response | 0 | 0 | 0 | 1 | 3
  No response | 4 | 2 | 1 | 1 | 11
  Not reported | 1 | 0 | 0 | 0 | 0
  Response Undetermined | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Who Died, Serious Adverse Events (SAEs), Adverse Events (AEs) and AEs Leading to Study Drug Discontinuation
Description: AE: New untoward medical occurrence or worsening of a preexisting medical condition that does not have causal relationship with this treatment. SAE: Untoward medical event that at any dose: results in death, persistent or significant disability/incapacity, drug dependency/abuse; life-threatening, an important medical event, a congenital anomaly/birth defect; requires inpatient hospitalization/prolongs existing hospitalization. Grade 1= Mild; Grade 2= Moderate; Grade 3= Severe; Grade 4 = Life-threatening or disabling.
Time Frame: Baseline (pretreatment), from the date of first dose until at least 30 days after the last dose of study drug (median duration of dasatinib treatment=5.2 months [range 0 to 33 months]).
Population: All treated participants, participants who received at least 1 dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 17
participants
  All deaths | 3 | 2 | 0 | 1 | 3
  Deaths within 30 days of last dose | 1 | 1 | 0 | 0 | 2
  All SAEs | 3 | 2 | 2 | 5 | 9
  Drug-related SAEs | 1 | 1 | 1 | 1 | 4
  AEs leading to discontinuation | 2 | 1 | 1 | 1 | 8
  Drug-related AEs leading to discontinuation | 2 | 0 | 0 | 0 | 7
  All AEs | 6 | 3 | 3 | 6 | 17
  Drug-related AEs | 6 | 3 | 3 | 6 | 17

6. Primary Outcome: Number of Participants With Hematology Abnormalities (Worst On-study Grade vs Baseline): Leukopenia, Neutropenia, Thrombocytopenia, and Anemia
Description: As per NCI CTCAE Version 3.0 criteria. Grade (GR)1=Mild; GR2=Moderate; GR3=Severe; GR4=Life-threatening or disabling. White blood cell (WBC):GR1=<LLN(lower limit of normal)-3.0*10^9/L; GR2=<3.0-2.0*10^9/L; GR3:<2.0-1.0*10^9/L; GR4:<1.0*10^9/L. LLN=lower limit of normal. Absolute Neutrophil Count (ANC): GR1=<LLN-1.5*10^9/L; GR2=<1.5-1.0*10^9/L; GR3:<1.0-0.5*10^9/L; GR4:<0.5*10^9/L. Hemoglobin: GR1=<LLN-10.0g/dL; GR2=<10.0-8.0g/dL; GR3:<8.0-6.5g/dL; GR4:<6.5g/dL. Platelets: GR1=<LLN-75.0*10^9/L; GR2=<75.0-50.0*10^9/L; GR3:<50.0-25.0*10^9/L; GR4:<25.0*10^9/L. BL=Baseline; PBL=post baseline.
Time Frame: Baseline (pretreatment); Cycles 1 and 2 (within 24 hours of Days 1, 4, 8, 11, 15, 18, 21, and 25); beyond Cycle 2 (within 24 hours of Days 1 and 15,off treatment visit ) (median duration of dasatinib treatment=5.2 mo [range 0 to 33 mo])
Population: All treated participants, participants who received at least 1 dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 17
participants
  Leukopenia; GR 0 at BL, GR 0 PBL | 0 | 2 | 0 | 1 | 2
  Leukopenia; GR 0 at BL, GR 1 to 2 PBL | 1 | 1 | 3 | 2 | 6
  Leukopenia; GR 0 at BL, GR 3 to 4 PBL | 2 | 0 | 0 | 0 | 3
  Leukopenia; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  Leukopenia; GR 1 to 2 at BL, GR 1 to 2 PBL | 0 | 0 | 0 | 0 | 1
  Leukopenia; GR 1 to 2 at BL, GR 3 to 4 PBL | 3 | 0 | 0 | 3 | 5
  Neutropenia; GR 0 at BL, GR 0 PBL | 0 | 1 | 0 | 0 | 1
  Neutropenia; GR 0 at BL, GR 1 to 2 PBL | 2 | 1 | 2 | 3 | 3
  Neutropenia; GR 0 at BL, GR 3 to 4 PBL | 3 | 1 | 1 | 0 | 8
  Neutropenia; GR 1 to 2 at BL, GR 0 | 0 | 0 | 0 | 0 | 0
  Neutropenia; GR 1 to 2 at BL, GR 1 to 2 PBL | 0 | 0 | 0 | 0 | 1
  Neutropenia; GR 1 to 2 at BL, GR 3 to 4 PBL | 1 | 0 | 0 | 3 | 4
  Thrombocytopenia; GR 0 at BL, GR 0 PBL | 0 | 1 | 0 | 1 | 2
  Thrombocytopenia; GR 0 at BL, GR 1 to 2 PBL | 3 | 1 | 2 | 3 | 5
  Thrombocytopenia; GR 0 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 2
  Thrombocytopenia; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  Thrombocytopenia; GR 1 to 2 at BL, GR 1 to 2 PBL | 1 | 0 | 1 | 1 | 3
  Thrombocytopenia; GR 1 to 2 at BL, GR 3 to 4 PBL | 2 | 1 | 0 | 1 | 5
  Anemia; GR 0 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  Anemia; GR 0 at BL, GR 1 to 2 PBL | 0 | 1 | 1 | 3 | 6
  Anemia; GR 0 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 1
  Anemia; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  Anemia; GR 1 to 2 at BL, GR 1 to 2 PBL | 4 | 1 | 1 | 1 | 5
  Anemia; GR 1 to 2 at BL, GR 3 to 4 PBL | 1 | 1 | 1 | 1 | 5
  Anemia; GR 3 to 4 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  Anemia; GR 3 to 4 at BL, GR 1 to 2 PBL | 0 | 0 | 0 | 0 | 0
  Anemia; GR 3 to 4 at BL, GR 3 to 4 PBL | 1 | 0 | 0 | 0 | 0
  Anemia; GR Not reported at BL | 0 | 0 | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Serum Chemistry Abnormalities (Worst On-study Grade vs Baseline): Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Total Bilirubin (TB), and Serum Creatinine (SC)
Description: Grading as per NCI CTCAE Version 3.0 criteria. GR1=Mild; GR2=Moderate; GR3=Severe; GR4=Life-threatening or disabling. Aspartate aminotransferase (AST) and alanine aminotransferase(ALT): GR1=>ULN-2.5*ULN (upper limit of normal); GR2=>2.5-5.0*ULN; GR3=>5.0-20.0*ULN; GR4:>20.0*ULN; TB:GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3-10*ULN, GR4=>10*ULN; SC: GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3.0-6.0*ULN, GR4=>6.0*ULN. BL=Baseline; PBL=post baseline.
Time Frame: as for outcome 6
Population: All treated participants, participants who received at least 1 dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 17
participants
  AST; GR 0 at BL, GR 0 PBL | 4 | 0 | 2 | 5 | 5
  AST; GR 0 at BL, GR 1 to 2 PBL | 2 | 2 | 0 | 0 | 8
  AST; GR 0 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 0
  AST; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  AST; GR 1 to 2 at BL, GR 1 to 2 PBL | 0 | 1 | 1 | 1 | 3
  AST; GR 1 to 2 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 1
  High ALT; GR 0 at BL, GR 0 PBL | 2 | 1 | 1 | 2 | 5
  ALT; GR 0 at BL, GR 1 to 2 PBL | 4 | 0 | 0 | 3 | 9
  ALT; GR 0 at BL, GR 3 to 4 PBL | 0 | 1 | 1 | 0 | 0
  ALT; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  ALT; GR 1 to 2 at BL, GR 1 to 2 PBL | 0 | 1 | 1 | 1 | 2
  ALT; GR 1 to 2 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 1
  Total Bilirubin; GR 0 at BL, GR 0 PBL | 5 | 1 | 2 | 4 | 13
  Total Bilirubin; GR 0 at BL, GR 1 to 2 PBL | 1 | 1 | 1 | 2 | 4
  Total Bilirubin; GR 0 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 0
  SC; GR 0 at BL, GR 0 PBL | 4 | 1 | 1 | 6 | 12
  SC; GR 0 at BL, GR 1 to 2 PBL | 2 | 1 | 2 | 0 | 3
  SC; GR 0 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 1
  SC; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  SC; GR 1 to 2 at BL, GR 1 to 2 PBL | 0 | 1 | 0 | 0 | 0
  SC; GR 1 to 2 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 1

8. Secondary Outcome: Number of Participants With Partial Response
Description: Partial response was achieved when there was ≥50% reduction of serum M-protein (Mpr)and reduction in 24 hour urinary Mpr by ≥90% or to <200 mg/24 hr. If the serum and urine Mpr were unmeasurable, a ≥50% decrease in the difference between involved and uninvolved free light chain (FLC) levels was required in place of the Mpr criteria. If serum, urine Mpr, and serum FLC assay were unmeasurable, ≥50% reduction in plasma cells was required in place of Mpr, provided baseline bone marrow plasma cell percentage was ≥30%; a ≥50% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: Baseline, at the end of the treatment period (median duration of dasatinib treatment=5.2 months [range 0 to 33 months]).
Population: All treated participants, participants who received at least 1 dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 17
participants | 1 | 1 | 2 | 4 | 3

9. Secondary Outcome: Number of Participants With Minimal Response
Description: Response criteria was based on The International Uniform Response Criteria for Multiple Myeloma (with a slight modification). Minimal Response was achieved when there was 25% to 49% reduction of serum M-Protein, 50% to 89% reduction in 24 hour urinary M-protein which still exceeded 200 mg/24 hour. If the serum and urine M-protein were unmeasurable, 25% to 49% reduction in plasma cells was required. In addition, if present at baseline, a 25% to 49% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: Baseline, at the end of the treatment period (median duration of dasatinib treatment=5.2 months [range 0 to 33 months]).
Population: All treated participants, participants who received at least 1 dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 17
participants | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Serum Chemistry Abnormalities (Worst On-study Grade vs Baseline): High Calcium, Low Calcium, Low Magnesium, and Low Phosphorus
Description: Grading as per NCI CTCAE Version 3.0 criteria. GR1=Mild; GR2=Moderate; GR3=Severe; GR4=Life-threatening or disabling. Calcium (low): GR1: <LLN - 8.0 mg/dL, GR2: <8.0 - 7.0 mg/dL, GR3: <7.0 - 6.0 mg/dL, GR4: <6.0 mg/dL. Calcium (High): GR1: >ULN - 11.5 mg/dL, GR2: >11.5 - 12.5 mg/dL, GR3: >12.5 - 13.5 mg/dL, GR4: >13.5 mg/dL. Magnesium (Low): GR1: <LLN - 1.2 mg/dL, GR2: <1.2 - 0.9 mg/dL, GR3: <0.9 - 0.7 mg/dL, GR4: <0.7 mg/dL. Phosphorus (low): GR1: <LLN - 2.5 mg/dL, GR2: <2.5 - 2.0 mg/dL, GR3: <2.0 - 1.0 mg/dL, GR4: <1.0 mg/dL. BL=Baseline; PBL=post baseline.
Time Frame: as for outcome 6
Population: All treated participants, participants who received at least 1 dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg
Number analyzed (Participants) | 6 | 3 | 3 | 6 | 17
participants
  High Calcium; GR 0 at BL, GR 0PBL | 4 | 2 | 3 | 4 | 15
  High Calcium; GR 0 at BL, GR 1 to 2 PBL | 1 | 0 | 0 | 0 | 1
  High Calcium; GR 0 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 0
  High Calcium; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  High Calcium; GR 1 to 2 at BL, GR 1 to 2 PBL | 0 | 1 | 0 | 2 | 1
  High Calcium; GR 1 to 2 at BL, GR 3 to 4 PBL | 1 | 0 | 0 | 0 | 0
  Low Calcium; GR 0 at BL, GR 0 PBL | 2 | 0 | 1 | 2 | 1
  Low Calcium; GR 0 at BL, GR 1 to 2 PBL | 3 | 2 | 2 | 4 | 12
  Low Calcium; GR 0 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 2
  Low Calcium; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  Low Calcium; GR 1 to 2 at BL, GR 1 to 2 PBL | 1 | 1 | 0 | 0 | 1
  Low Calcium; GR 1 to 2 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 1
  Low Magnesium; GR 0 at BL, GR 0 PBL | 2 | 1 | 3 | 2 | 7
  Low Magnesium; GR 0 at BL, GR 1 to 2 PBL | 3 | 2 | 0 | 3 | 6
  Low Magnesium; GR 0 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 1
  Low Magnesium; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  Low Magnesium; GR 1 to 2 at BL, GR 1 to 2 PBL | 1 | 0 | 0 | 1 | 3
  Low Magnesium; GR 1 to 2 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 0
  Low Magnesium; GR Not reported at BL | 0 | 0 | 0 | 0 | 0
  Low Phosphorus; GR 0 at BL, GR 0 PBL | 1 | 0 | 2 | 3 | 8
  Low Phosphorus; GR 0 at BL, GR 1 to 2 PBL | 3 | 3 | 0 | 2 | 2
  Low Phosphorus; GR 0 at BL, GR 3 to 4 PBL | 1 | 0 | 0 | 1 | 6
  Low Phosphorus; GR 1 to 2 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  Low Phosphorus; GR 1 to 2 at BL, GR 1 to 2 PBL | 0 | 0 | 0 | 0 | 0
  Low Phosphorus; GR 1 to 2 at BL, GR 3 to 4 PBL | 0 | 0 | 0 | 0 | 1
  Low Phosphorus; GR 3 to 4 at BL, GR 0 PBL | 0 | 0 | 0 | 0 | 0
  Low Phosphorus; GR 3 to 4 at BL, GR 1 to 2 PBL | 0 | 0 | 0 | 0 | 0
  Low Phosphorus; GR 3 to 4 at BL, GR 3 to 4 PBL | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg
Serious Adverse Events (participants affected / at risk) | 2/3 | 5/6 | 9/17 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 17/17 | 0/6 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg (N=3) | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (N=6) | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (N=17) | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg (N=6) | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg (N=3)
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 4 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0
Blood viscosity increased (Investigations) | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 100 mg + Lenalidomide 20 mg + Dexamethasone 40 mg (N=3) | Dasatinib 100 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (N=6) | Dasatinib 140 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (N=17) | Dasatinib 70 mg + Lenalidomide 15 mg + Dexamethasone 40 mg (N=6) | Dasatinib 70 mg + Lenalidomide 20 mg + Dexamethasone 40 mg (N=3)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 8 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 4 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 7 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 3 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 4 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 4 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 5 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 2 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 3 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 8 | 0 | 0
Crying (General disorders) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Dysacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Effusion (General disorders) | 0 | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 6 | 0 | 0
IIIrd nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 4 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 9 | 0 | 0
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 6 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 3 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 3 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Anger (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 12 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 14 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 8 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 6 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 10 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 10 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.